CLINICAL TRIAL: NCT07211412
Title: Effects of Acute Cryotherapy on Musculoskeletal Function and Biomarkers for Inflammation, Oxidative Stress, and Muscle Damage
Brief Title: Acute Cryotherapy on Musculoskeletal Function and Biomarkers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Responsible Party: Principal Investigator, Alvaro Gurovich, Professor and Chair, University of Texas, El Paso
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2356825
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Exercise Induced Muscle Damage; Cryotherapy
Keywords: Exercise induced muscle damage; Cryotherapy; Cold-pack; Ice-pack; Eccentric exercise; Creatine kinase; c-reactive protein; interlukin-6; 8-isoprostane; Range of motion; Maximal Voluntary Isometric Contraction; Pain
MeSH Terms: conditions — Pain | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, controlled clinical trial with 3 independent groups.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control-control (No Intervention): This arm will include no intervention and only functional assessments and blood draws for biomarkers.
- Control (Placebo Comparator): This arm will have eccentric exercise-induced muscle damage on day 0 and then 15-min of room temperature cold-pack immediately after and then for 4 more days every 24 hours.
  Interventions: Other: Eccentric exercise-induced muscle damage
- Cryotherapy (Active Comparator): This arm will have eccentric exercise-induced muscle damage on day 0 and then 15-min of cold (-5°C) cold-pack immediately after and then for 4 more days every 24 hours.
  Interventions: Other: Cryotherapy; Other: Eccentric exercise-induced muscle damage

INTERVENTIONS:
Other: Cryotherapy — A cold (-5°C) cold-pack for 15 minutes every 24 hours for 5 days
  Other Names: cold-pack; ice-pack
  Arms: Cryotherapy
Other: Eccentric exercise-induced muscle damage — 3 sets of 15 repetitions of eccentric contractions at 80% of 1RM. This is to induced a controlled muscle damage in 2 of the 3 arms.
  Other Names: doms
  Arms: Control; Cryotherapy

SUMMARY:
In 2020, Dubois and Esculier proposed a paradigm shift in the acute management of musculoskeletal injuries, advocating for the transition from the traditional PRICE protocol- Protect, Rest, Ice, Compression, Elevation-to the more holistic PEACE & LOVE framework. This updated model emphasizes Protection, Elevation, Avoiding anti-inflammatories, Compression, and Education, followed by Load, Optimism, Vascularization, and Exercise. Notably, the PEACE & LOVE approach omits the use of ice, a decision that has sparked considerable debate. While the rationale centers on avoiding interference with the natural inflammatory and regenerative processes, this omission stands in contrast to a substantial body of animal research suggesting that cryotherapy can mitigate secondary tissue injury by reducing inflammation and metabolic activity. Despite its widespread clinical use, human studies have yet to provide conclusive evidence supporting or refuting the efficacy of cryotherapy in acute injury management, leaving clinicians to navigate between tradition, emerging evidence, and evolving philosophies of care. Even though it is important to consider natural inflammation for a better regenerative process, animal models have shown that the original injury can elicit oxidative stress, which will enhance cellular damage (secondary damage) and inflammation. Clinically, it is unknown if this secondary damage would increase functional impairment.

Therefore, this proposal will determine if cryotherapy can decrease secondary damage, after exercise-induced muscle damage, and if this decrease is associated to lower inflammation, oxidative stress and functional impairments.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, controlled clinical trial with 3 independent groups. One group (control-control or CON-CON) will not exercise and will not have any cryotherapy intervention, a second group (control or CON) will exercise but use a "room temperature" cold-pack, and the cryotherapy group (CRYO) will exercise and receive a cold cold-pack every day for 15-min.

We anticipate to compare means in several markers (functional and in blood) using a two-way analysis of variance (ANOVA, time x condition) where time is before, and 0, 24, 48, 72, 96, and 264 hours after exercise (6 visits) and conditions are CON-CON, CON, and CRYO.

VISIT ONE Before the informed consent process, potential participants will rest for 10 minutes, and their blood pressure will be taken to confirm eligibility. Once eligibility is confirmed, participants will go through the informed consent process. After the participants have signed the informed consent, the participants will be randomly allocated to one of the 3 groups. Then, a blood sample (two 10-ml tubes) from an antecubital vein of the dominant arm will be drawn. After the blood drawn, a set of functional tests ( i.e., arm girth, active range of motion (ROM), peak pressure threshold (PPT), and maximal voluntary isometric contraction (MVIC)) will be performed (the description of each test can be found below). Once the functional tests are performed, participants from the CON-CON group will be dismissed. Participants from the other 2 groups will perform a controlled exercise-induced muscle damage (EIMD) through eccentric exercise (protocol description below). Immediately after the EIMD protocol, participants in the CON group will receive 15-min of a room temperature cold-pack in room RSC 100. Participants in the CRYO group will receive 15-min of a cold cold-pack in room RSC 100. Treatment will be performed by RAs that were not involved in any testing session. After treatment, CON or CRYO, the same set of functional tests will be performed in room RSC 117.

VISIT TWO to FOUR (24, 48, and 72 hours after VISIT 1, respectively) Participants will get a blood draw (two 10-ml tubes) from an antecubital vein of the dominant arm. Then, participants in the CON group will receive 15-min of a room temperature cold-pack in room RSC 100. Participants in the CRYO group will receive 15-min of a cold cold-pack in room RSC 100. Treatment will be performed by RAs that were not involved in any testing session. Participants from the CON-CON group will not have any treatment. Finally, the set of functional tests will be performed.

VISIT FIVE (96 hours after VISIT 1) Participants will get only a blood draw (two 10-ml tubes) from an antecubital vein of the dominant arm. Then, participants in the CON group will receive 15-min of a room temperature cold-pack in room RSC 100. Participants in the CRYO group will receive 15-min of a cold cold-pack in room RSC 100. Treatment will be performed by RAs that were not involved in any testing session. Participants from the CON-CON group will not have any treatment.

VISIT SIX (264 hours after VISIT 1) Participants will get a blood draw (two 10-ml tubes) from an antecubital vein of the dominant arm. Then, the set of functional tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy
* normotensive
* non-smokers (all tobacco products including e-cigarettes)

Exclusion Criteria:

* Cardiovascular diseases (including hypertension)
* pregnancy
* any musculoskeletal injury 6 months prior the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Maximal Voluntary Isometric Contraction (MVIC) | From enrollment to the end of study at 12 days
  Laid down on an isokinetic dynamometer system (Humac-Norm, Computer Sports Medicine, inc., Stoughton, MA), participants will be asked to flex their non-dominant arm (pull with their hand) against the dynamometer. They will perform 3 tries with 1 minute between tries and the peak value will be considered the MVIC.
Peak Pressure Threshold (PPT) | From enrollment to the end of study at 12 days.
  PPT is the application of an algometer, which measure pressure on a specific body point (see figure below), while asking the participant 2 questions: 1) tell me when the pressure becomes pain and 2) how much pain you felt from 0 to 100, where 0 is no pain and 100 is the larger pain you have ever experienced. PPT will be performed over the flexor muscles (biceps brachialis) of the non-dominant arm.
Creatine kinase | From enrollment to the end of treatment at 5 days
  Blood biomarker of muscle damage. Blood draws will be performed before and 0, 24, 48, 72, and 96 hours after EIMD.
Interleukin-6 | From enrollment to the end of treatment at 5 days
  Blood biomarker of inflammation. Blood draws will be performed before and 0, 24, 48, 72, and 96 hours after EIMD.
8-isoprostane | From enrollment to the end of treatment at 5 days
  Blood biomarker of oxidative stress. Blood draws will be performed before and 0, 24, 48, 72, and 96 hours after EIMD.

SECONDARY OUTCOMES:
Arm girth | From enrollment to the end of study at 12 days.
  With a flexible tape measure, we will measure the perimeter of the non-dominant arm, on the middle between the shoulder and the elbow.
Active Range of Motion (ROM) | From enrollment to the end of study at 12 days.
  Participants will be asked to flex and extend the non-dominant elbow while wearing a wireless range of motion device (electronic goniometer, ActiveForce2, ActiveBody, San Diego, CA) (see picture below). The device will measure the active ROM.
C-reactive protein | From enrollment to the end of treatment at 5 days.
  Blood biomarker of inflammation. Blood draws will be performed before and 0, 24, 48, 72, and 96 hours after EIMD.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at El Paso, Rehabilitation Sciences Complex, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No
I might share un-identified data when submitting manuscripts, if asked to do so.

REFERENCES:
- [Background] Qu C, Wu Z, Xu M, Qin F, Dong Y, Wang Z, Zhao J. Cryotherapy Models and Timing-Sequence Recovery of Exercise-Induced Muscle Damage in Middle- and Long-Distance Runners. J Athl Train. 2020 Apr;55(4):329-335. doi: 10.4085/1062-6050-529-18. Epub 2020 Mar 11. PMID 32160058
- [Background] Pooley S, Spendiff O, Allen M, Moir HJ. Comparative efficacy of active recovery and cold water immersion as post-match recovery interventions in elite youth soccer. J Sports Sci. 2020 Jun-Jun;38(11-12):1423-1431. doi: 10.1080/02640414.2019.1660448. Epub 2019 Aug 28. PMID 31456474
- [Background] Rose C, Edwards KM, Siegler J, Graham K, Caillaud C. Whole-body Cryotherapy as a Recovery Technique after Exercise: A Review of the Literature. Int J Sports Med. 2017 Dec;38(14):1049-1060. doi: 10.1055/s-0043-114861. Epub 2017 Nov 21. PMID 29161748
- [Background] Kwiecien SY, McHugh MP, Hicks KM, Keane KM, Howatson G. Prolonging the duration of cooling does not enhance recovery following a marathon. Scand J Med Sci Sports. 2021 Jan;31(1):21-29. doi: 10.1111/sms.13822. Epub 2020 Sep 25. PMID 32901996
- [Background] Sasaki R, Sakamoto J, Kondo Y, Oga S, Takeshita I, Honda Y, Kataoka H, Origuchi T, Okita M. Effects of Cryotherapy Applied at Different Temperatures on Inflammatory Pain During the Acute Phase of Arthritis in Rats. Phys Ther. 2021 Feb 4;101(2):pzaa211. doi: 10.1093/ptj/pzaa211. PMID 33351944
- [Background] Merrick MA, Rankin JM, Andres FA, Hinman CL. A preliminary examination of cryotherapy and secondary injury in skeletal muscle. Med Sci Sports Exerc. 1999 Nov;31(11):1516-21. doi: 10.1097/00005768-199911000-00004. PMID 10589851
- [Background] Allan R, Malone J, Alexander J, Vorajee S, Ihsan M, Gregson W, Kwiecien S, Mawhinney C. Cold for centuries: a brief history of cryotherapies to improve health, injury and post-exercise recovery. Eur J Appl Physiol. 2022 May;122(5):1153-1162. doi: 10.1007/s00421-022-04915-5. Epub 2022 Feb 23. PMID 35195747
- [Background] Kwiecien SY, McHugh MP. The cold truth: the role of cryotherapy in the treatment of injury and recovery from exercise. Eur J Appl Physiol. 2021 Aug;121(8):2125-2142. doi: 10.1007/s00421-021-04683-8. Epub 2021 Apr 20. PMID 33877402
- [Background] Dubois B, Esculier JF. Soft-tissue injuries simply need PEACE and LOVE. Br J Sports Med. 2020 Jan;54(2):72-73. doi: 10.1136/bjsports-2019-101253. Epub 2019 Aug 3. No abstract available. PMID 31377722